CLINICAL TRIAL: NCT01576705
Title: Efficacy Assessment of Systematic Treatment With Folinic Acid and Thyroid Hormone on Psychomotor Development of Down Syndrome Young Children
Acronym: ACTHYF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Institut Jerome Lejeune (Other)
Collaborators: Hôpital Cochin (Other); Central Hospital, Nancy, France (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IJL-AFHT-TH10
Record Dates: First submitted 2012-04-11; First posted 2012-04-12 (Estimated); Results first posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2019-12

CONDITIONS: Down Syndrome
Keywords: Down syndrome; Young children; Psychomotor development; Thyroid hormone; Folinic acid; Psychometric tests; GMDS; Griffiths; Genetic factors; Biochemical factors
MeSH Terms: conditions — Down Syndrome | interventions — Thyroid Hormones; Leucovorin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Thyroxin + folinic acid (Experimental)
  Interventions: Drug: thyroid hormone and folinic acid
- Thyroxin+folinic acid placebo (Active Comparator)
  Interventions: Drug: thyroid hormone and folinic acid
- Thyroxin placebo+ folinic acid (Active Comparator)
  Interventions: Drug: thyroid hormone and folinic acid
- Thyroxin placebo+ folinic acid placebo (Placebo Comparator)
  Interventions: Drug: thyroid hormone and folinic acid

INTERVENTIONS:
Drug: thyroid hormone and folinic acid — thyroid hormone 25microg or placebo in tablets folinic acid 5 mg or placebo in capsules

SUMMARY:
Evaluation of the following in very young children with Down syndrome:

* the efficacy of systematic treatment with L-thyroxine at controlled doses (clinically and by ultrasensitive thyreostimulating hormone (TSH) assay),
* the efficacy of systematic folinic acid treatment at a dose of 1 mg/kg/o.i.d,
* any interaction between these two treatments.

ELIGIBILITY:
Inclusion Criteria:

* patient with a karyotype demonstrating homogeneous, free or Robertsonian translocation trisomy 21
* patient having undergone a cardiac ultrasound not demonstrating any severe heart disease
* patient aged 6 to 18 months at inclusion

Exclusion Criteria:

* congenital hypothyroidism
* hypothyroidism demonstrated by laboratory tests (TSH > 7mUI/l)
* presenting or having presented hyperthyroidism
* presenting or having presented leukaemia
* presenting or having presented West syndrome or any other form of epilepsy or unstable neurological disease
* presenting or having presented signs of central nervous system distress: stroke, postoperative hypoxia, meningitis)
* presenting severe heart disease on cardiac ultrasound, with haemodynamic effects
* presenting non-controlled cardiac arrhythmia
* Apgar < 7 to 5 min at birth
* Gestational age < 231 days (33 gestation weeks)

Ages: 6 Months to 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 175 (Actual)
Dates: Start 2012-04-02 (Actual); Primary Completion 2017-12-14 (Actual); Study Completion 2017-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clotilde MIRCHER, MD, Principal Investigator — Institut Jerome Lejeune, Paris, France; Franck STURTZ, MD, PhD, Study Chair — Department of Biochemistry and Molecular Genetics, Limoges University, Limoges, France
Locations (1):
- Institut Jerome Lejeune, Paris, France

REFERENCES:
- [Background] Blehaut H, Mircher C, Ravel A, Conte M, de Portzamparc V, Poret G, de Kermadec FH, Rethore MO, Sturtz FG. Effect of leucovorin (folinic acid) on the developmental quotient of children with Down's syndrome (trisomy 21) and influence of thyroid status. PLoS One. 2010 Jan 11;5(1):e8394. doi: 10.1371/journal.pone.0008394. PMID 20084109
- [Background] van Trotsenburg AS, Kempers MJ, Endert E, Tijssen JG, de Vijlder JJ, Vulsma T. Trisomy 21 causes persistent congenital hypothyroidism presumably of thyroidal origin. Thyroid. 2006 Jul;16(7):671-80. doi: 10.1089/thy.2006.16.671. PMID 16889491
- [Background] van Trotsenburg AS, Vulsma T, van Rozenburg-Marres SL, van Baar AL, Ridder JC, Heymans HS, Tijssen JG, de Vijlder JJ. The effect of thyroxine treatment started in the neonatal period on development and growth of two-year-old Down syndrome children: a randomized clinical trial. J Clin Endocrinol Metab. 2005 Jun;90(6):3304-11. doi: 10.1210/jc.2005-0130. Epub 2005 Mar 8. PMID 15755847
- [Background] Ellis JM, Tan HK, Gilbert RE, Muller DP, Henley W, Moy R, Pumphrey R, Ani C, Davies S, Edwards V, Green H, Salt A, Logan S. Supplementation with antioxidants and folinic acid for children with Down's syndrome: randomised controlled trial. BMJ. 2008 Mar 15;336(7644):594-7. doi: 10.1136/bmj.39465.544028.AE. Epub 2008 Feb 21. PMID 18296460
- [Derived] Sacco S, Bouis C, Gallard J, Pichot A, Blondiaux E, Marey I, Dorison N, Sturtz F, Cieuta-Walti C, Ravel A, Mircher C. Psychomotor development in infants and young children with Down syndrome-A prospective, repeated measure, post-hoc analysis. Am J Med Genet A. 2022 Mar;188(3):818-827. doi: 10.1002/ajmg.a.62587. Epub 2021 Dec 4. PMID 34863019
- [Derived] Mircher C, Sacco S, Bouis C, Gallard J, Pichot A, Le Galloudec E, Cieuta C, Marey I, Greiner-Mahler O, Dorison N, Gambarini A, Stora S, Durand S, Polak M, Baruchel A, Schlumberger E, Dewailly J, Azar-Kolakez A, Gueant-Rodriguez RM, Gueant JL, Borderie D, Bonnefont-Rousselot D, Blondiaux E, Ravel A, Sturtz FG. Thyroid hormone and folinic acid in young children with Down syndrome: the phase 3 ACTHYF trial. Genet Med. 2020 Jan;22(1):44-52. doi: 10.1038/s41436-019-0597-8. Epub 2019 Jul 8. PMID 31281181
- See also: Institut Jerome Lejeune — http://www.institutlejeune.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment period : 2012-2016 First inclusion : 02/04/2012 Last inclusion : 14/12/2016
  Location : Institut Jérôme Lejeune
Pre-assignment Details: As recruitment was nationwide and patients were included at a single centre, screening and randomisation were performed on the same day to minimise visits to the centre. Eligibility of randomised patients for TSH levels per exclusion criterion #8 was thus confirmed retrospectively, and patients with high TSH levels were discontinued.
Groups:
- Thyroxin + Folinic Acid: thyroid hormone and folinic acid: thyroid hormone 25microg in tablets folinic acid 5 mg in capsules
- Thyroxin+Folinic Acid Placebo: thyroid hormone and folinic acid: thyroid hormone 25microg in tablets folinic acid placebo in capsules
- Thyroxin Placebo+ Folinic Acid: thyroid hormone and folinic acid: thyroid hormone placebo in tablets folinic acid 5 mg in capsules
- Thyroxin Placebo+ Folinic Acid Placebo: thyroid hormone and folinic acid: thyroid hormone placebo in tablets folinic acid placebo in capsules
Period: Overall Study
Arm/Group | Thyroxin + Folinic Acid | Thyroxin+Folinic Acid Placebo | Thyroxin Placebo+ Folinic Acid | Thyroxin Placebo+ Folinic Acid Placebo
Started | 43 | 45 | 43 | 44
Completed | 40 | 37 | 38 | 41
Not Completed | 3 | 8 | 5 | 3
Not completed — TSH > 7 mIU/L at baseline | 3 | 7 | 5 | 3
Not completed — invalid ICF | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: The modified intention-to-treat (mITT) population included all randomized patients who did not prematurely discontinue due to elevated baseline thyroid stimulating hormone (TSH)
Groups:
- Total: Total of all reporting groups
Arm/Group | Thyroxin + Folinic Acid | Thyroxin+Folinic Acid Placebo | Thyroxin Placebo+ Folinic Acid | Thyroxin Placebo+ Folinic Acid Placebo | Total
Number analyzed (Participants) | 40 | 37 | 38 | 41 | 156
Age, Customized [Mean (Standard Deviation); unit: months] — Age at inclusion in months
  months
    Age | 12.3 (3.4) | 12.2 (3.8) | 12.3 (4) | 12.7 (3.3) | 12.37 (3.58)
Sex: Female, Male [Count of Participants; unit: Participants] — Male or Female
  Participants
    Female | 17 | 16 | 17 | 17 | 67
    Male | 23 | 21 | 21 | 24 | 89
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  France | 40 | 37 | 38 | 41 | 156
Patient's height at baseline [Mean (Standard Deviation); unit: cm] — Height measured in cm
  cm | 70.86 (3.88) | 71.14 (5.03) | 71.13 (4.15) | 71.68 (4.36) | 71.21 (4.33)
Karyotype % [Count of Participants; unit: Participants]
  Free trisomy 21 | 39 | 37 | 38 | 40 | 154
  Robertsonian translocation | 1 | 0 | 0 | 1 | 2
Pregnancy term [Mean (Standard Deviation); unit: weeks of amenorrhea] | 38.03 (1.37) | 38.14 (0.98) | 38.29 (1.33) | 37.85 (0.99) | 38.07 (1.18)
Cardiac abnormalities [Number; unit: participants]
  Isolated hear murmur | 1 | 3 | 2 | 1 | 7
  Atrioventricular septal defect (AVSD) | 2 | 1 | 1 | 2 | 6
TSH [Mean (Standard Deviation); unit: mIU/L] | 4.3 (1.7) | 4.32 (1.52) | 4.79 (1.23) | 4.45 (1.49) | 4.46 (1.5)
Patient's weight at baseline [Mean (Standard Deviation); unit: Kg] — Weight measured in kg
  Kg | 8.30 (1.2) | 8.19 (1.42) | 8.54 (1.13) | 8.62 (1.6) | 8.42 (1.35)
Patient's head circumference at baseline [Mean (Standard Deviation); unit: cm] — Head circumference measured in cm
  cm | 43.5 (1.59) | 43.55 (1.64) | 43.63 (1.55) | 43.82 (1.68) | 43.63 (1.6)

OUTCOME MEASURES:

1. Primary Outcome: GMDS (Griffiths Mental Development Scale)
Description: GMDS for testing and estimate babies psychomotor development from birth to 2 years trough six subscales : Locomotor, Personal-social, Hearing and language, Eye-Hand coordination, Performance.Sub- and General Quotients (GDQ) standard score are based on a mean of 100 and a standard deviation of 16. For children with delayed development, which is the case for children with Down Syndrome, Quotient tables could be not used because sub- and General quotient floors at 50. For each subscale, a raw score was derived from the contributing items. Total raw score was obtained by adding subscale raw scores. Sum of all subscale raw scores was converted into a development age using correspondence table. Subscale and global development quotients were computed by dividing the development age by the chronological age multiplied by 100. For preterm infants, chronological age was corrected taking into account the gestational term. Higher QD's scores show a better psychomotor development outcome
Time Frame: 12 months
Population: The main analysis of the primary efficacy endpoint is the adjusted change from baseline in GDQ derived from the Griffith Mental Development Scales (GMDS) at 12 months analysed by ANCOVA adjusted for covariates. Expected Outcome : six points difference in GDQ between any of the three treatment group compared to placebo at 12 months from baseline.
Measure: Mean (Standard Deviation); unit: developpement quotient
Arm/Group | Thyroxin + Folinic Acid | Thyroxin+Folinic Acid Placebo | Thyroxin Placebo+ Folinic Acid | Thyroxin Placebo+ Folinic Acid Placebo
Number analyzed (Participants) | 38 | 35 | 30 | 41
developpement quotient | 51.96 (7.88) | 51.27 (6.48) | 51.66 (6.37) | 51.67 (8.29)

2. Secondary Outcome: BL (Brunet Lezine Revised Scale)
Description: BL includes 4 subscales : Locomotor, Coordination, Language, Sociability. Subscale and global developpemental quotients were computed by dividing the developpemental age by the chronological age multiplied by 100. This kind of formula do not give a min-max outcome. Higher QD's scores show a better psychomotor developpement outcome.
Time Frame: 12 months
Population: The main analysis of the secondary efficacy endpoint of the adjusted change from baseline in the BL-R GDQ at 12 months, analysed by ANCOVA adjusted for covariates, is presented in the mITT population.
Measure: Mean (Standard Deviation); unit: developpement quotient
Arm/Group | Thyroxin + Folinic Acid | Thyroxin+Folinic Acid Placebo | Thyroxin Placebo+ Folinic Acid | Thyroxin Placebo+ Folinic Acid Placebo
Number analyzed (Participants) | 38 | 35 | 30 | 40
developpement quotient | 51.18 (6.98) | 50.64 (7.25) | 51.24 (6.46) | 51.36 (8.27)

ADVERSE EVENTS:
Time Frame: 12 months
Description: safety analysis were performed on all randomised patients receiving at least one dose of study treatment Safety population correspond to 174 subjects
Arm/Group | Thyroxin+Folinic Acid Placebo | Thyroxin + Folinic Acid | Thyroxin Placebo+ Folinic Acid | Thyroxin Placebo+ Folinic Acid Placebo
All-Cause Mortality (participants affected / at risk) | 0/44 | 1/43 | 0/43 | 0/44
Serious Adverse Events (participants affected / at risk) | 9/44 | 8/43 | 8/43 | 5/44
Other Adverse Events (participants affected / at risk) | 0/44 | 0/43 | 7/43 | 0/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thyroxin+Folinic Acid Placebo (N=44) | Thyroxin + Folinic Acid (N=43) | Thyroxin Placebo+ Folinic Acid (N=43) | Thyroxin Placebo+ Folinic Acid Placebo (N=44)
Infections and infestations (Infections and infestations) | 3 (3) | 4 (4) | 2 (2) | 5 (7)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 4 (5) | 4 (6) | 3 (5) | 0 (0)
General disorders and administration site conditions (General disorders) | 0 (0) | 2 (2) | 1 (1) | 0 (0)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 2 (3) | 0 (0) | 0 (0) | 1 (1)
Surgical and medical procedures (Surgical and medical procedures) | 2 (2) | 0 (0) | 1 (1) | 0 (0)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Neoplasm begign, maligant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Skin and subcutnaeous tissue disorders (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Thyroxin+Folinic Acid Placebo (N=44) | Thyroxin + Folinic Acid (N=43) | Thyroxin Placebo+ Folinic Acid (N=43) | Thyroxin Placebo+ Folinic Acid Placebo (N=44)
Endocrine disorders (Endocrine disorders) | 0 (0) | 0 (0) | 5 (5) | 0 (0)
Neoplasms begnin, malignant and unspecified (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nervous system disorders (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
The initial protocol planned for 256 patients, however due to difficulties in recruiting patients, the sample size was subsequently reduced to 175 patients, to obtain 140 evaluable patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-11-07): https://cdn.clinicaltrials.gov/large-docs/05/NCT01576705/Prot_SAP_000.pdf